CLINICAL TRIAL: NCT00258388
Title: A Randomized Phase II Study of OGX-011 in Combination With Docetaxel and Prednisone or Docetaxel and Prednisone Alone in Patients With Metastatic Hormone Refractory Prostate Cancer
Brief Title: Docetaxel and Prednisone With/Out OGX-011 in Recurrent or Metastatic Prostate Cancer That Did Not Respond to Previous Hormone Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I165; CAN-NCIC-IND165 (Other: PDQ); ONCOGENEX-OGX-011-03 (Other: Oncogenex Technologies); FHCRC-6084 (Other: Fred Hutchinson Cancer Research Center); UWCC-UW-6084 (Other: University of Washington); UWCC-06-0499-H/D (Other: University of Washington); CDR0000450846 (Other: PDQ)
Record Dates: First submitted 2005-11-22; First posted 2005-11-24 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2020-04

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; recurrent prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- OGX011, Docetaxel and Prednisone (Active Comparator)
  Interventions: Drug: custirsen sodium; Drug: docetaxel; Drug: prednisone
- Docetaxel plus prednisone (Active Comparator)
  Interventions: Drug: docetaxel; Drug: prednisone

INTERVENTIONS:
Drug: custirsen sodium — 640mg IV for 2 hours - Cycle 1: Days -7, -5, -3, 1, 8, 15 (4 week cycle)
  Subsequent cycles:
  weekly on days 1, 8, 15 (3 week cycles)
  Arms: OGX011, Docetaxel and Prednisone
Drug: docetaxel — 75mg/m2 IV for 1 hour - Day 1 every 3 weeks (3 week cycles)
Drug: prednisone — 5mg PO BID

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel and prednisone, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. OGX-011 may help docetaxel and prednisone kill more tumor cells by making tumor cells less resistant to the drugs.

PURPOSE: This randomized phase II trial is studying how well giving docetaxel and prednisone with or without OGX-011 works in treating patients with recurrent or metastatic prostate cancer that did not respond to previous hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy, in terms of prostate-specific antigen response, of docetaxel and prednisone with or without OGX-011 in patients with hormone-refractory locally recurrent or metastatic prostate cancer.

Secondary

* Determine the objective response rate and duration in patients treated with these regimens.
* Determine the safety and toxic effects of these regimens in these patients.
* Determine the overall and progression-free survival of patients treated with these regimens.

OUTLINE: This is a multicenter, randomized, open-label study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive a loading dose of OGX-011 IV over 2 hours on days -7, -5, and -3. Patients then receive OGX-011 IV over 2 hours on days 1, 8, and 15, docetaxel IV over 1 hour on day 1, and oral prednisone twice daily on days 1-21. Treatment repeats every 3 weeks for up to 10 courses in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive docetaxel IV over 1 hour on day 1 and oral prednisone twice daily on days 1-21. Treatment repeats every 3 weeks for up to 10 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 80 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the prostate

  * Metastatic or locally recurrent disease
* Not curable with standard therapy
* Systemic chemotherapy is indicated, due to disease progression while receiving androgen-ablative therapy (i.e., hormone-refractory disease)

  * Disease progression is defined as development of new metastatic lesions OR ≥ 2 consecutive rises in prostate-specific antigen (PSA) over a reference value
  * Androgen ablative therapy must have included either medical or surgical castration

    * Castrate level of testosterone (≤ 1.7 nmol/L) required if treated with medical androgen ablation
  * Patients with documented disease progression while on peripheral antiandrogens must also have documented PSA progression after stopping antiandrogens
* PSA ≥ 5 ng/mL
* No known CNS metastases

PATIENT CHARACTERISTICS:

Performance status

* ECOG 0-2

Life expectancy

* At least 12 weeks

Hematopoietic

* Absolute granulocyte count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* No known bleeding disorder

Hepatic

* PT and PTT or INR normal
* Bilirubin normal
* AST and ALT ≤ 1.5 times upper limit of normal (ULN)

Renal

* Creatinine ≤ 1.5 times ULN

Cardiovascular

* No significant cardiac dysfunction

Other

* Fertile patients must use effective contraception
* No pre-existing peripheral neuropathy ≥ grade 2
* No active, uncontrolled infection
* No significant neurological disorder that would preclude study compliance
* No history of other malignancies within the past 5 years except adequately treated nonmelanoma skin cancer

PRIOR CONCURRENT THERAPY:

Chemotherapy

* No prior chemotherapy except estramustine and recovered
* No other concurrent chemotherapy

Endocrine therapy

* See Disease Characteristics
* At least 4 weeks since prior antiandrogens (6 weeks for bicalutamide)
* Luteinizing hormone-releasing hormone (LHRH) agonist therapy must be continued* or restarted* during study treatment to maintain castrate levels of testosterone NOTE: *For patients receiving LHRH agonist therapy prior to study entry

Radiotherapy

* At least 4 weeks since prior external beam radiotherapy except low-dose, nonmyelosuppressive radiotherapy

  * Must have had less than 25% of marrow irradiated
* No prior strontium chloride Sr 89
* No concurrent radiotherapy except low-dose, nonmyelosuppressive, palliative radiotherapy

Surgery

* At least 2 weeks since prior major surgery

Other

* At least 4 weeks since prior investigational agent
* At least 4 weeks since prior anticancer therapy
* No concurrent therapeutic anticoagulants except low-dose oral anticoagulants (i.e., 1 mg warfarin) or low molecular weight heparin
* No other concurrent investigational agents
* No other concurrent cytotoxic therapy

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2005-09-28 (Actual); Primary Completion 2007-11-08 (Actual); Study Completion 2011-01-18 (Actual)

PRIMARY OUTCOMES:
Prostate-specific antigen (PSA) response measured by Bubley criteria at completion of study | 2 years

SECONDARY OUTCOMES:
Toxicity | 2 years
Time to treatment failure | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Kim N. Chi, MD, Study Chair — British Columbia Cancer Agency
Locations (13):
- University of Washington, Seattle, Washington, United States
- Canada (12):
  - Tom Baker Cancer Centre, Calgary
  - Cross Cancer Institute, Edmonton
  - QEII Health Sciences Center, Halifax
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton
  - BCCA - Cancer Centre for the Southern Interior, Kelowna
  - London Regional Cancer Program, London
  - CHUM - Hopital Notre-Dame, Montreal
  - Atlantic Health Sciences Corporation, Saint John
  - Odette Cancer Centre, Toronto
  - Univ. Health Network-Princess Margaret Hospital, Toronto
  - BCCA - Vancouver Cancer Centre, Vancouver
  - CancerCare Manitoba, Winnipeg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chi KN, Hotte SJ, Yu EY, Tu D, Eigl BJ, Tannock I, Saad F, North S, Powers J, Gleave ME, Eisenhauer EA. Randomized phase II study of docetaxel and prednisone with or without OGX-011 in patients with metastatic castration-resistant prostate cancer. J Clin Oncol. 2010 Sep 20;28(27):4247-54. doi: 10.1200/JCO.2009.26.8771. Epub 2010 Aug 23. PMID 20733135